CLINICAL TRIAL: NCT00003160
Title: A Phase II Trial of Paclitaxel (Taxol) Administered as a Weekly One Hour Infusion in Patients With Taxol/Platinum-Refractory Stage III and IV Ovarian Cancer
Brief Title: Weekly Infusions of Paclitaxel in Treating Women With Stage III or Stage IV Ovarian Cancer Refractory to Paclitaxel and Platinum
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Theradex (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000065955; THERADEX-B97-3250; BMS-TAX/MEN.03; NCI-V97-1366
Record Dates: First submitted 1999-11-01; First posted 2004-05-27 (Estimated); Last update posted 2011-04-20 (Estimated); Status verified 2001-01

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; recurrent ovarian epithelial cancer; fallopian tube cancer; primary peritoneal cavity cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Paclitaxel

INTERVENTIONS:
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Giving the drugs in different ways may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of paclitaxel in treating women with stage III or stage IV ovarian cancer that is refractory to paclitaxel and platinum-based regimens.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the objective response rate of paclitaxel given as a weekly one hour infusion in patients with paclitaxel/platinum refractory stage III and IV ovarian cancer. II. Evaluate the safety of paclitaxel in this patient population. III. Assess the overall survival in these patients. IV. Assess quality of life in these patients.

OUTLINE: This is a multicenter, open label, nonrandomized study. Patients are administered paclitaxel as a one hour IV infusion every 7 days. Each cycle consists of four weeks. Treatment may be delayed for up to 2 weeks and there is no limit to the number of interruptions a patient may experience. Patients receive paclitaxel weekly until disease progression or unacceptable toxicity. Treatment is assessed every 3 cycles for one year and then every 6 months thereafter during study. Quality of life is assessed every cycle for the first 6 cycles, then every 3 cycles thereafter. Patients are followed every 3 months for survival.

PROJECTED ACCRUAL: There will be 100 patients accrued into this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed stage III or IV ovarian cancer that is refractory to an initial chemotherapy regimen that included a platinum agent plus paclitaxel - Epithelial ovarian cancer - Primary carcinoma of the peritoneum - Fallopian tube cancer Initial response to platinum and paclitaxel must have been one of the following: Progression or stable disease Response that lasted less than 3 months Response that lasted at least 3 months, but when retreated with both agents (in combination or as single agents) disease was refractory Measurable or evaluable disease Evaluable disease is defined by: CA-125 at least 100 units/mL AND CA-125 level must have at least doubled from baseline determination

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: At least 3 months Hematopoietic: Absolute granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 2 times upper limit of normal (ULN) AST or ALT no greater than 2.5 times ULN Renal: Creatinine no greater than 2.0 mg/dL Cardiovascular: No New York Heart Association Class III or IV heart disease No myocardial infarction within last 6 months No congestive heart failure No unstable angina No clinically significant pericardial effusion or arrhythmia Neurology: No current peripheral neuropathy of any etiology that is greater than grade 1 Other: No active serious infection or other serious underlying medical condition No prior significant allergic reactions to drugs containing Cremophor, such as teniposide, cyclosporin, or vitamin K Not pregnant or nursing Adequate contraception required of all fertile patients

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 3 weeks since immunotherapy No concurrent immunotherapy Chemotherapy: Prior paclitaxel treatment must have been administered on a 3 week or greater schedule No other prior chemotherapy besides platinum and paclitaxel At least 3 weeks since acceptable chemotherapy Endocrine therapy: At least 3 weeks since hormonal therapy No concurrent hormonal therapy Radiotherapy: At least 3 weeks since radiotherapy No prior radiation to greater than 30% of bone marrow Surgery: At least 3 weeks since major surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 1997-09

CONTACTS AND LOCATIONS:
Overall Officials: Maurie Markman, MD, Study Chair — The Cleveland Clinic
Locations (18):
- United States (18):
  - Oncology Center at Providence Park, Mobile, Alabama
  - Hematology Associates, Ltd., Phoenix, Arizona
  - Highlands Oncology Group, P.A., Fayetteville, Arkansas
  - Cancer Center of Santa Barbara, Santa Barbara, California
  - Good Samaritan Medical Center, West Palm Beach, Florida
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Creighton University Cancer Center, Omaha, Nebraska
  - Jersey Shore Cancer Center, Neptune City, New Jersey
  - Women's Health Center at Albany Medical Center, Albany, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Akron General Medical Center, Akron, Ohio
  - Oncology/Hematology Care, Inc., Cincinnati, Ohio
  - Cleveland Clinic Cancer Center, Cleveland, Ohio
  - Women's Cancer Center of Central PA, P.C., Harrisburg, Pennsylvania
  - Women and Infants Hospital of Rhode Island, Providence, Rhode Island
  - Brookview Research, Inc., Nashville, Tennessee
  - Harrington Cancer Center, Amarillo, Texas
  - Rockwood Clinic P.S., Spokane, Washington